CLINICAL TRIAL: NCT02415803
Title: Safety and Efficacy of Low-Dose Ticagrelor in Chinese Patients With Non-ST-Elevation Acute Coronary Syndrome: A Randomized Clinical Trial
Brief Title: Safety and Efficacy of Low-Dose Ticagrelor in Chinese Patients With NSTE-ACS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACS-1
Record Dates: First submitted 2015-03-26; First posted 2015-04-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2014-12

CONDITIONS: Non ST Segment Elevation Acute Coronary Syndrome
Keywords: low-dose ticagrelor; clopidogrel; Chinese patients with NSTE-ACS; platelet reactivity; inhibition of platelet aggregation
MeSH Terms: interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- low-dose ticagrelor (Experimental): To observe the safety and efficacy of low-dose ticagrelor in Chinese patients with non-ST-elevation acute coronary syndrome
  Interventions: Drug: low-dose ticagrelor
- conventional-dose ticagrelor (Active Comparator): To observe the different safety and efficacy between low-dose ticagrelor and conventional-dose ticagrelor.
  Interventions: Drug: conventional-dose ticagrelor
- clopidogrel (Active Comparator): To observe the different safety and efficacy between low-dose ticagrelor and conventional-dose clopidogrel.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: low-dose ticagrelor — 90 mg loading dose, then 45 mg twice daily for 5 days
  Arms: low-dose ticagrelor
Drug: conventional-dose ticagrelor — 180 mg loading dose, then 90 mg twice daily for 5 days
  Arms: conventional-dose ticagrelor
Drug: Clopidogrel — 300 mg loading dose, then 75 mg once daily for 5 days
  Arms: clopidogrel

SUMMARY:
Ticagrelor is an oral, reversibly-binding, direct-acting P2Y12 receptor antagonist used clinically for the prevention of atherothrombotic events in patients with acute coronary syndromes (ACS). Guideline recommendations on the use of dual antiplatelet therapy (DAPT) have been formulated that ticagrelor 90 mg twice daily plus aspirin in preference to clopidogrel 75mg daily plus aspirin for patients who have an ACS with or without ST-segment elevation. These recommendations are primarily based on large, randomized, Phase III clinical trials. However, few East Asian patients (or those of East Asian descent) have been included in these trials to assess the use of these drugs. In addition, a growing body of data supported that East Asian might have different adverse event profiles (thrombophilia and bleeding) and "therapeutic window" compared with white subjects. Furthermore, "East Asian paradox" phenomenon has been described that East Asian patients have a higher prevalence of platelet reactivity during DAPT, but an ischaemic event rate following PCI or ACS is similar or even lower than white patients. Therefore, the antiplatelet treatment strategy that is most appropriate for East Asian patients is increasingly urgent. Therefore, we performed the current study to observe the different effects of low-dose ticagrelor (45 mg twice daily), conventional-dose ticagrelor (90 mg twice daily) and clopidogrel (75mg once daily) on high platelet reactivity (HPR) and IPA, and investigated the safety and efficacy of low-dose ticagrelor further in Chinese patients with non-ST-elevation ACS (NSTE-ACS).

DETAILED DESCRIPTION:
Ticagrelor is an oral, reversibly-binding, direct-acting P2Y12 receptor antagonist used clinically for the prevention of atherothrombotic events in patients with acute coronary syndromes (ACS). Guideline recommendations on the use of dual antiplatelet therapy (DAPT) have been formulated that ticagrelor 90 mg twice daily plus aspirin in preference to clopidogrel 75mg daily plus aspirin for patients who have an ACS with or without ST-segment elevation. These recommendations are primarily based on large, randomized, Phase III clinical trials. However, few East Asian patients (or those of East Asian descent) have been included in these trials to assess the use of these drugs. In addition, a growing body of data supported that East Asian might have different adverse event profiles (thrombophilia and bleeding) and "therapeutic window" compared with white subjects. Furthermore, "East Asian paradox" phenomenon has been described that East Asian patients have a higher prevalence of platelet reactivity during DAPT, but an ischaemic event rate following PCI or ACS is similar or even lower than white patients. Therefore, the antiplatelet treatment strategy that is most appropriate for East Asian patients is increasingly urgent. In Korea and Japan, it has been reported that low doses of ticagrelor had a more potent inhibition of platelet aggregation (IPA) than clopidogrel (75 mg once daily) in healthy subjects and patients with stable coronary artery disease, respectively. But it is still not clear whether a low dose of ticagrelor is superior to clopidogrel in a large population of Chinese ACS patients. A recent study on pharmacokinetics and tolerability of ticagrelor has found that maximum plasma concentration (Cmax) and area under the plasma concentration-time curve (AUC) of ticagrelor (90 mg twice daily) and its active metabolite (AR-C124910XX) tended to be approximately 40% higher in healthy Chinese volunteers compared with Caucasian subjects. This data also suggested that a low dose of ticagrelor might be more appropriate for Chinese ACS patients. In view of a large diurnal variation with a single daily dose, a lower dose twice daily may be a better choice for Chinese patients. Therefore, we performed the current study to observe the different effects of low-dose ticagrelor (45 mg twice daily), conventional-dose ticagrelor (90 mg twice daily) and clopidogrel (75mg once daily) on high platelet reactivity (HPR) and IPA, and investigated the safety and efficacy of low-dose ticagrelor further in Chinese patients with non-ST-elevation ACS (NSTE-ACS).

ELIGIBILITY:
Inclusion Criteria:

* hospitalized for NSTE-ACS within the preceding 48 h
* have one of the following additional criteria:

  1. ischemic symptoms at rest, lasting ≥10 minutes;
  2. horizontal or down-sloping ST segment depression ≥0.1 mV;
  3. cardiac troponin I (cTnI), marker associated with NSTE-ACS, local laboratory upper limit of normal values;
  4. underwent percutaneous coronary intervention (PCI); (5) a history of myocardial infarction.

Exclusion Criteria:

* ST-elevation ACS;
* planned use of glycoprotein IIb/IIIa receptor inhibitors, adenosine diphosphate (ADP) receptor antagonists, or anticoagulant therapy during the study period;
* platelet count <100g/L;
* creatinine clearance rate < 30ml/min;
* diagnosed as respiratory or circulatory instability (cardiac shock, severe congestive heart failure NYHA II-IV or left ventricular ejection fraction < 40%);
* a history of bleeding tendency;
* aspirin, ticagrelor or clopidogrel allergies;
* diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the differences in mean inhibition of platelet aggregation or inhibition ratio (%) | before dosing (baseline) and up to 12 hours after the last dose
  After overnight fasting, venous blood samples of all subjects were taken for pharmacodynamic measurements before dosing (baseline) and 12 hours after the last dose. VerifyNow P2Y12 (Accumetrics, SanDiego, CA), a whole-blood, cartridge-based and point-of-care turbidometric assay, was performed to test platelet aggregation at baseline and 12 hours after the last dose, and the results were reported in P2Y12 reaction units (PRU). With this assay, a higher PRU reflects greater adenosine-diphosphate-mediated platelet reactivity (PR). High-platelet reactivity (HPR) was defined as a PRU>208. Blood samples were placed in 3.2% sodium citrate (Greiner Bio-One Vacuette North America, Inc, Monroe, NC) for this assay. Additionally, inhibition of platelet aggregation (IPA) calculated by VerifyNow assays was similar to light transmittance aggregometry.

SECONDARY OUTCOMES:
Number of bleeding events | throughout the study (from baseline to 12 hours after the last dose)
Number of difficulty breathing events | throughout the study (from baseline to 12 hours after the last dose)
number of ventricular pauses | throughout the study (from baseline to 12 hours after the last dose)
number of myocardial infarction events | throughout the study (from baseline to 12 hours after the last dose)
number of death events | throughout the study (from baseline to 12 hours after the last dose)
number of stroke events | throughout the study (from baseline to 12 hours after the last dose)
number of severe recurrent ischemia events | throughout the study (from baseline to 12 hours after the last dose)

CONTACTS AND LOCATIONS:
Locations (1):
- VerifyNow, San Diego, California, United States